CLINICAL TRIAL: NCT02014506
Title: Haploidentical Allogeneic Hematopoietic Stem Cell Transplantation in Children and Adolescents
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ho Joon Im, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCPHO-SCT1303
Record Dates: First submitted 2013-12-04; First posted 2013-12-18 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Haploidentical Hematopoietic Stem Cell Transplantation; Malignant Disease; Non-malignant Disease
Keywords: Children and adolescents; Malignant disease; Non-malignant disease; TCRαβ depletion; Haploidentical hematopoietic stem cell transplantation
MeSH Terms: interventions — fludarabine; Cyclophosphamide; Antilymphocyte Serum; Filgrastim; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAPLO (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: anti-thymocyte globulin; Biological: filgrastim; Radiation: Total body irradiation; Procedure: TCRαβ-depleted hematopoietic cell transplantation; Device: CliniMACS

INTERVENTIONS:
Drug: Fludarabine — 40mg/M2 once daily IV on days -7 to -2
Drug: Cyclophosphamide — 50 mg/kg IV on day -3 and -2
Biological: anti-thymocyte globulin
Biological: filgrastim — Beginning on day 4 and continuing until blood counts recover
Radiation: Total body irradiation — 200 cGy per day on D-6 to -4 (eligible disease except aplastic anemia) 200 cGy per day on D-5 & -4 (severe aplastic anemia)
Procedure: TCRαβ-depleted hematopoietic cell transplantation
Device: CliniMACS — Immunogenetic depletion of TCRαβ cells

SUMMARY:
Purpose of study: This phase I/II trial is to evaluate the safety and feasibility of TCRαβ-depleted graft from haploidentical family donors in treating children and adolescents with malignant or non-malignant diseases.

ELIGIBILITY:
Inclusion Criteria:

A. Disease inclusions

1. Hematologic malignancy:

   * Acute lymphoblastic leukemia including induction failure, CR1 (Ph+, t(4:11), hypodiploid and other very high risk features), ≥ CR2, infant ALL with MLL or other unfavorable features
   * Acute myeloid leukemia excluding CR1 with t(8:21), inv(16), t(15:17), and Down syndrome
   * Myelodysplastic syndrome: RCC with -7 or RCC in need of transfusion
   * Chronic myeloid leukemia in AP
   * Juvenile myelomonocytic leukemia
   * Malignant lymphoma, NHL or HD, after failed autologous HSCT
   * Other
2. Non-hematologic malignancy

   * Relapsed or refractory solid tumors including neuroblastoma, rhabdomyosarcoma and so on
3. Non-malignant hematologic disease

   * Acquired severe and very severe aplastic anemia
   * Fanconi anemia
   * Paroxysmal nocturnal hemoglobinuria
   * Congenital dyserythropoietic anemia
   * Others
4. Inherited or metabolic disease

   * Hemophagocytic lymphohistiocytosis
   * Malignant osteopetrosis
   * Storage diseases
   * Others B. Recipient inclusions

1. Age < 21 years 2. No HLA-identical stem cell donor available 3. Lansky-Play performance score >60 4. No active infection at the time of transplantation

Exclusion Criteria:

1. HIV-infection
2. Presence of active and serious infection
3. Cardiac ejection fraction <35% on echocardiography
4. Severe pulmonary dysfunction (DLCO <30%)
5. Liver function abnormalities with bilirubin >4mg/dL and elevation of transaminases > 400U/L
6. Concurrent severe or uncontrolled medical disease
7. Patients who are pregnant
8. Patients unwilling or unable to comply with the protocol or unable to give informed consent

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate tralsplant-related mortality after haploidentical hematopoietic stem cell transplantation using TCRαβ-depleted graft | 1 year posttransplant

SECONDARY OUTCOMES:
To assess engraftment and graft failure | 28 days posttransplant
To estimate the risk of acute GVHD | 100 days posttransplant
To estimate the incidence of relapse | 100 days and 1 year post-transplant
To estimate the incidence and severity of chronic GVHD | 1 year posttransplant
To estimate the overall survival | 1 year posttransplant
To estimate the incidence of bacterial, fungal and viral infection | 100 days and 1 year posttransplant
To estimate the reactivation rate of CMV, EBV | 100 days and 1 year posttransplant
To evaluate the immune reconstitution of T, B, and NK cells | days 7, 14, 21, 28, 60, 90, 180, 270, and 365 days post-transplant
To evaluate the lineage-specific chimerism using flow cytomery of CD3+, CD19, CD56, TCR αβ, and TCRγδ at pre-transplant | days 7, 10, 14, 21, 28, 60, 90, 180, 270 and 365 post-transplant
To assess event free survival | 1 year posttransplant

CONTACTS AND LOCATIONS:
Overall Officials: Ho Joon Im, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Park JA, Koh KN, Choi ES, Jang S, Kwon SW, Park CJ, Seo JJ, Im HJ. Successful rescue of early graft failure in pediatric patients using T-cell-depleted haploidentical hematopoietic SCT. Bone Marrow Transplant. 2014 Feb;49(2):270-5. doi: 10.1038/bmt.2013.163. Epub 2013 Oct 21. PMID 24141651
- [Background] Im HJ, Koh KN, Choi ES, Jang S, Kwon SW, Park CJ, Chi HS, Seo JJ. Excellent outcome of haploidentical hematopoietic stem cell transplantation in children and adolescents with acquired severe aplastic anemia. Biol Blood Marrow Transplant. 2013 May;19(5):754-9. doi: 10.1016/j.bbmt.2013.01.023. Epub 2013 Feb 1. PMID 23380343
- [Background] Schumm M, Lang P, Bethge W, Faul C, Feuchtinger T, Pfeiffer M, Vogel W, Huppert V, Handgretinger R. Depletion of T-cell receptor alpha/beta and CD19 positive cells from apheresis products with the CliniMACS device. Cytotherapy. 2013 Oct;15(10):1253-8. doi: 10.1016/j.jcyt.2013.05.014. PMID 23993299
- See also: Stem cell transplant — http://www.mayoclinic.com/health/stem-cell-transplant/MY00089/METHOD=print
- See also: fludarabine — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a692003.html
- See also: cyclophosphamide — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a682080.html
- See also: leukemia — http://www.nlm.nih.gov/medlineplus/leukemia.html